CLINICAL TRIAL: NCT05654896
Title: Prophylactic Antibiotic Use in Transarterial Chemoembolization for Hepatocellular Carcinoma: an Open-label, Randomised, Prospective Study
Brief Title: Prophylactic Antibiotic Use in Transarterial Chemoembolization for Hepatocellular Carcinoma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nadeem Iqbal (Other)
Collaborators: Ahmad Zia (Unknown); Muhammad Junaid Tahir (Unknown)
Responsible Party: Sponsor-Investigator, Nadeem Iqbal, PakistanKidney, Pakistan Kidney and Liver Institute and Research Center
Organization: Pakistan Kidney and Liver Institute and Research Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PKLI-IRB/AP/89
Record Dates: First submitted 2022-12-08; First posted 2022-12-16 (Actual); Last update posted 2022-12-16 (Actual); Status verified 2022-12

CONDITIONS: Antibiotic Prophylaxis
Keywords: Antibiotic; TACE; HCC
MeSH Terms: interventions — Ceftriaxone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No Antibiotic Prophylaxis Group (No Intervention): No antibiotic will be administered prophylactically for TACE.
- Antibiotic Prophylaxis Group (Experimental): Antibiotic will be administered prophylactically (i.e., Inj. Ceftriaxone 1g, intravenous × stat)
  Interventions: Drug: Ceftriaxone Sodium

INTERVENTIONS:
Drug: Ceftriaxone Sodium — Antibiotic will be administered prophylactically for TACE
  Arms: Antibiotic Prophylaxis Group

SUMMARY:
This study aims to determine the effectiveness of prophylactic antibiotic use for TACE and occurrence of postoperative liver abscess.

There would be two comparison groups. Current standard of care treatment at PKLI&RC (as per local guidelines) would be given to all patients receiving TACE for the intervention group or 'antibiotic group' (i.e., Inj. Ceftriaxone 1g, intravenous × stat). While no antibiotic would be given to the 'no antibiotic group'.

DETAILED DESCRIPTION:
Liver cancer especially hepatocellular carcinoma (HCC) is among the top five most common carcinomas in the world. According to the latest Cardiovascular and Interventional Radiological Society of Europe (CIRSE) standards of practice guidelines (2021), routine antibiotic prophylaxis is not recommended. However, prophylactic antibiotics are recommended in cases where there is a high risk of developing a liver abscess. These include biliary obstruction or the presence of a bilioenteric anastomosis. This study aims to determine the effectiveness of prophylactic antibiotic use for TACE and occurrence of postoperative liver abscess.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of primary liver cancer or hepatocellular carcinoma.
2. Patients receiving TACE in PKLI & RC.
3. Patients giving informed consent.

Exclusion Criteria:

1. Receiving two or more TACE during the same hospitalization
2. Use of any antibiotics other than the prophylactic antibiotic in 48hours prior to TACE
3. Known hypersensitivity to specified antibiotic used in the study
4. Incomplete or missing laboratory investigations and data
5. Taking Sorafenib before TACE
6. TACE combined with ablation or immunetherapy
7. Tumor size >10 cm
8. Portal vein thrombosis
9. Dilated biliary channels on CT scan / Billiary invasion by tumor

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Estimated)
Dates: Start 2022-11-26 (Actual); Primary Completion 2023-11-26 (Estimated); Study Completion 2023-12-26 (Estimated)

PRIMARY OUTCOMES:
Leukocytosis | 2 days
  Predominantly neutrophilic leukocytosis ( > 11 ×109/L) with fever ( > 38 °C) in upto 48 hours post-TACE
Liver abscess | 30 days
  Occurrence of liver abscess as diagnosed by imaging within 30 days of the procedure
Liver abscess and intervention | 30 days
  Liver abscess requiring an intervention (e.g., percutaneous transhepatic abscess drainage (PTAD), percutaneous transhepatic abscess puncture or liver abscess incision) within 30 days of TACE

CONTACTS AND LOCATIONS:
Overall Officials: Ahmad Zia Ud Din, Principal Investigator — PKLI & RC, Lahore
Locations (1):
- Pakistan Kidney and Liver Institute, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-12-05): https://cdn.clinicaltrials.gov/large-docs/96/NCT05654896/Prot_SAP_000.pdf